CLINICAL TRIAL: NCT00046800
Title: A Randomized, Open Label Phase II Study of OSI-211 vs Topotecan in Patients With Advanced and/or Recurrent Epithelial Ovarian Cancer
Brief Title: Study of OSI-211 vs. Topotecan in Patients With Relapsed Epithelial Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 110-20
Record Dates: First submitted 2002-10-03; First posted 2002-10-04 (Estimated); Last update posted 2011-10-20 (Estimated); Status verified 2011-10

CONDITIONS: Ovarian Neoplasms
Keywords: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — lurtotecan

INTERVENTIONS:
Drug: OSI-211 (Liposomal Lurtotecan)

SUMMARY:
The purpose of this study is to estimate the efficacy and safety of OSI-211 and topotecan in patients with relapsed epithelial ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed relapsed ovarian cancer.
* Measurable disease greater than or equal to 20 mm (or greater than or equal to 10 mm on spiral CT scan).
* One or two prior regimens of chemotherapy. At least one regimen must have contained cisplatin or carboplatin.
* At least three weeks since prior chemotherapy and recovery from any related toxicities.
* At least four weeks since prior radiotherapy and recovery from any related toxicities.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2002-09; Study Completion 2003-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (2):
  - NYU- Kaplan Comprehensive Cancer Center, New York, New York
  - The Sarah Cannon Cancer Center, Centennial Medical Center, Nashville, Tennessee
- United Kingdom (9):
  - St Chad's Unit, Birmingham
  - Beatson Oncology Centre, Glasgow
  - Royal Surrey County Hospital, Guildford, Surrey
  - Royal Marsden NHS Trust, London
  - Northern Centre for Cancer Research, Newcastle General Hospital, Newcastle upon Tyne
  - Mount Vernon Hospital, Northwood, Middlesex
  - CRC Department of Medical Oncology, Sutton Surrey
  - Taunton & Somerset Hospital, Taunton
  - Medical Oncology Unit, Torbay District General Hospital, Torquay